CLINICAL TRIAL: NCT07179133
Title: Additional Effects of Semispinalis Cervicis Strengthening With Craniocervical Flexion Training on Chronic Neck Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2025/02
Record Dates: First submitted 2025-09-11; First posted 2025-09-17 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Chronic Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Craniocervical Flexion Training (Active Comparator): Detailed components of Craniocervical Flexion (CCF) Training
  Interventions: Procedure: Craniocervical Flexion Training alone
- Semispinalis Cervicis Strengthening with CCF Training (Active Comparator): Detailed components of Semispinalis Cervicis Strengthening and Craniocervical Flexion (CCF) Training
  Interventions: Procedure: Semispinalis Cervicis strengthening with Craniocervical Flexion Training:

INTERVENTIONS:
Procedure: Craniocervical Flexion Training alone — 10-minute hot pack treatment before starting the protocol. Week 1: Muscle Activation, • Hold for 5-10 seconds.
  * Perform in supine with a sphygmomanometer device.
  * Nod head gently as if saying "yes," aiming for 20-22 mmHg. Week 2: Endurance Training Goal: • Hold for 10-15 seconds. Increase holding time and precision.
  Exercise:
  • Maintain the contraction at 24-26 mmHg on the device. Week 3: Strength and Postural Training •Hold for 15 seconds.
  Exercise:
  * Perform CCFT in sitting or standing. Week 4: Functional Integration
  * Maintain contraction during functional tasks (e.g., desk work).
  * Hold for 15-20 seconds.
  * Sets/Reps: 3 sets of 8-12 repetitions.
  Arms: Craniocervical Flexion Training
Procedure: Semispinalis Cervicis strengthening with Craniocervical Flexion Training: — Craniocervical flexion training will be same as given to group A.
  Week 1: Semispinalis Cervicis Activation:
  * Patient sits upright with neutral spine.
  * Therapist applies gentle manual resistance at C2 vertebra while the patient resists backward motion.
  * Hold for 3-5 seconds, then relax.
  Week 2: Progressive Activation with Increased Resistance:
  * Apply moderate manual resistance at C2.
  * Hold for 5 seconds, focusing on controlled movement.
  Week 3: Strength and Functional Coordination with Dynamic Resistance:
  * Introduce light movement (e.g., slight backward head tilt) under resistance.
  * Therapist adjusts resistance dynamically.
  Week 4: Advanced Endurance and Functional Integration with Functional Movements:
  * Combine resistance training with controlled head rotations or slight lateral flexion.
  * Maintain resistance and stability.
  * Reps/Sets: 3-4 sets of 12 reps.
  Arms: Semispinalis Cervicis Strengthening with CCF Training

SUMMARY:
Chronic neck pain affects 30-50% of individuals annually and is a leading cause of disability, often linked to muscle imbalances and compensatory over activation of superficial muscles. While craniocervical flexion trainning (CCFT) improves neuromuscular control and reduces pain, limited researches has examined the additional benefits of semispinalis cervicis strengthening. This randomized controlled trial, conducted at Fauji Foundation Hospital and Foundation University College of Physical Therapy will assess the effects of combining semispinalis cervicis strengthening with CCFT on pain, cervical erange of motion, muscle strength and functional disability. Participants will be randomly assigned to either CCFT alone or CCFT with semispinalis cervicis strengthening, performed three times per week for four weeks. Data will be collected at baseline, mid study (week 2) and end of study (week 4) using the Numeric pain rating scale, Goniometer, Sphygmomanometer and Nexk disability index. This study addresses a research gap by exploring deep cervical extensors strengthening alongside CCFT, potentially improving rehabilitation strategies for pain relief, cervical stability and functional recovery.

DETAILED DESCRIPTION:
Detailed Description:

Chronic neck pain is persistent discomfort in the neck lasting over three months, often caused by poor posture, injury or degenerative conditions. It is the fourth-leading cause of disability worldwide, affecting 30-50% of people annually. Chronic neck pain significantly impacts quality of life, as well as physical and mental function, making it a leading cause of disability that is often challenging to manage. Common clinical symptoms include persistent neck pain, restricted neck movement, pain in the shoulders or upper limbs, migraines, muscle imbalances, and irregular breathing patterns. Chronic neck pain is often associated with a decline in the strength and endurance of deep neck muscles, particularly the deep cervical flexors (DCF) like the longus colli and longus capitis. These muscles are crucial for maintaining proper neck posture and stability. When they weaken, it can lead to poor posture and increased pain. Likewise deep neck flexors, deep cervical extensor muscles, which include the multifidus and semispinalis cervicis are also weakened in chronic neck pain patient's leading to increase pain and reduced ROMs. In response to the weakness of the deep neck muscles, the body activates superficial flexors and extensors to compensate for the loss of stability and strength. This compensatory activation is a natural response to maintain neck function and posture. However, relying on these superficial muscles can lead to over-activation, which is not ideal for long-term neck health. Exercise is essential for managing neck pain, with recent research highlighting the benefits of deep cervical muscle training. Craniocervical flexor exercises improve neuromuscular control, reduce pain, and enhance muscle activation. Likewise, deep cervical extensors like the semispinalis and multifidus play a key role in stabilization and should be targeted in rehabilitation.

Thavatchai et.al, conducted a study that shows Semispinalis cervicis strengthening outcomes benefits over usual-care outcomes for pain, cervical ROMs and functional disability.

Isha Sikka et al, conducted a study that Craniocervical Flexion training effectively reduces Neck Pain and improves functional status.

A study conducted by Ahmad H. Alghadir et.al, concluded that combining deep cervical flexor (DCF) training with conventional exercises significantly reduces pain and forward head posture (FHP) in school teachers.

Johannes Blomgren et.al, conducted a study found that applying manual resistance to the C2 vertebral arch resulted in the most selective activation of the semispinalis cervicis muscle (measured at C3) compared to resistance at the occiput or C5 level.

Jochen Schomacher et.al, concluded that targeting the semispinalis cervicis muscle through specific exercises, such as manual resistance in extension, can enhance its activation and potentially reduce neck pain.

Gorajiya et.al concludes that craniocervical flexion exercises are superior to isometric exercises, scapulothoracic exercises and transcutaneous electrical nerve stimulation alone in managing chronic neck pain.

Interventions Description:

Both groups will receive a 10-minute hot pack treatment before starting the protocol. Three sessions per week for 4 weeks.

Group A: Craniocervical Flexion Training protocol Group B: Semispinalis Cervicis strengthening in addition to the Craniocervical Flexion Training protocol.

Group A: Craniocervical Flexion Training alone

Week 1: Muscle Activation Goal:

Activate deep cervical flexors with the sphygmomanometer device.

Exercise:

* Perform in supine with a sphygmomanometer device.
* Nod head gently as if saying "yes," aiming for 20-22 mmHg.
* Hold for 5-10 seconds. Sets/Reps: 3 sets of 5 repetitions. Focus: Avoid activation of superficial neck muscles (e.g., sternocleidomastoid).

Week 2: Endurance Training Goal:

Increase holding time and precision.

Exercise:

* Maintain the contraction at 24-26 mmHg on the device.
* Hold for 10-15 seconds.
* Sets/Reps: 3 sets of 6-8 repetitions.

Week 3: Strength and Postural Training Goal:

Improve muscle strength and integrate postural control.

Exercise:

* Perform CCFT in sitting or standing.
* Progress to 28-30 mmHg and hold for 15 seconds.
* Sets/Reps: 3 sets of 8-10 repetitions.

Week 4: Functional Integration Goal:

Incorporate CCFT into daily activities.

Exercise:

* Maintain contraction during functional tasks (e.g., desk work).
* Hold for 15-20 seconds.
* Sets/Reps: 3 sets of 8-12 repetitions.

Group B: Semispinalis Cervicis strengthening with Craniocervical Flexion Training:

Craniocervical flexion training will be same as given to group A.

Week 1: Semispinalis Cervicis Activation:

* Patient sits upright with neutral spine.
* Therapist applies gentle manual resistance at C2 vertebra while the patient resists backward motion.
* Hold for 3-5 seconds, then relax.
* Reps/Sets: 2 sets of 6 reps. Focus: Avoid compensatory movements and maintain smooth activation

Week 2: Progressive Activation with Increased Resistance:

* Apply moderate manual resistance at C2.
* Hold for 5 seconds, focusing on controlled movement.
* Reps/Sets: 3 sets of 8 reps.
* Focus: Proper engagement of both semispinalis cervicis and deep cervical flexors.

Week 3: Strength and Functional Coordination with Dynamic Resistance:

* Introduce light movement (e.g., slight backward head tilt) under resistance.
* Therapist adjusts resistance dynamically. Reps/Sets: 3 sets of 10 reps

Week 4: Advanced Endurance and Functional Integration with Functional Movements:

* Combine resistance training with controlled head rotations or slight lateral flexion.
* Maintain resistance and stability.
* Reps/Sets: 3-4 sets of 12 reps. Focus: Smooth, coordinated and pain-free execution

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 35.
* Chronic nonspecific Neck Pain persisting for more than 3 months.
* Willingness to participate and and signed an informed consent form.
* Self reported neck pain intensity greater than and equal to 3 on 11 point numerical pain scale.

Exclusion Criteria:

* Recent neck injuries and surgeries.
* Several medical conditions like Hypertension, RA and Cardiovascular Diseases.
* Significant psychiatric disorders.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Chronic Neck Pain | 4 weeks
  Chronic Neck Pain will be measured using Numeric Pain Rating Scale, minimum value is 0 and maximum value is 10.
Neck Range of Motion | 4 weeks
  Neck Range of Motion will be measured using Goniometer, minimum and maximum value depends on movement.
Neck Muscle Strength | 4 weeks
  Neck Muscle Strength will be measured with Sphygmomanometer, minimum and maximm value depends on hold time of 20mmHg.
Neck Functional Disability | 4 weeks
  Neck Disability Index will be used to measure Neck Functional Disability, 0 to 50 is range.

CONTACTS AND LOCATIONS:
Overall Officials: Andleeb Zahra, Principal Investigator — Foundation University Islamabad
Locations (1):
- Foundation University Islamabad, Islamabad, Punjab Province, Pakistan